CLINICAL TRIAL: NCT01958853
Title: An Open Label Extension Trial for Patients With Fibromyalgia Who Complete Study NPT-201 (NCT01825954) and Who Experience Inadequate Pain Reduction
Brief Title: Prospective Evaluation of Reduced Impedance Noninvasive Cortical Electrostimulation (RINCE) to Reduce Fibromyalgia Effects - Extension Study
Acronym: PERRFECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cerephex Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPT-201E
Record Dates: First submitted 2013-10-04; First posted 2013-10-09 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-09

CONDITIONS: Fibromyalgia
Keywords: Pain
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 12-week RINCE (Experimental): RINCE - active RINCE therapy involving 24 total treatment applications from the NeuroPoint device
  Interventions: Device: RINCE

INTERVENTIONS:
Device: RINCE — The NeuroPoint device is used to deliver repeat applications of RINCE therapy
  Other Names: RINCE therapy; RINCE therapy using the NeuroPoint device

SUMMARY:
The purpose of this open label study is to provide up to 24 active treatments of noninvasive cortical electrostimulation therapy only to those fibromyalgia patients who experienced inadequate pain reduction in a sham controlled double blinded lead in study, NPT-201 (NCT01825954). The therapy will be provided by the NeuroPoint device using the same protocol as that used in active treatment arms of NPT-201. The study's primary outcome measure will be the patient's change from baseline in self-reported 24-hour average pain intensity. The study will provide active treatment to those participants who received sham therapy in NPT-201, and will test whether or not additional therapy applications might further improve pain in those participants who previously received active therapy, but did not achieve adequate pain relief.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have successfully completed study NPT-201 and had an inadequate pain response, defined as <50% reduction in pain from baseline during participation in NPT-201.
* Patient must provide written informed consent and privacy authorization prior to participation in the study.
* Female patients of childbearing potential must be willing to use an acceptable method of birth control for the duration of their study participation. Acceptable birth control includes a vasectomized partner, contraceptives (oral, parenteral, or transdermal), intrauterine device, or double barrier method including condoms, sponge, diaphragm, or vaginal ring with spermicidal jellies or cream. Patients considered not of childbearing potential must be surgically sterile (total hysterectomy, bilateral salpingo-oophorectomy, or tubal ligation) or greater than one year post-menopausal, defined as a complete cessation of menstruation for at least one year.
* Patients must be willing to refrain from all excluded therapies for the duration of the study.
* In the opinion of the Investigator, the patient is willing and able to comply with all protocol-specified requirements.

Exclusion Criteria:

* Patient has a current significant psychological or psychiatric disorder (e.g., severe, unstable or poorly controlled depression, severe anxiety or obsessive-compulsive disorder.
* Patient has a score of 2 or 3 on item 9 of the BDI, or, based on the investigator's judgment, the patient is at risk of suicidal ideation or behavior.
* Patient has resumed treatment with duloxetine, milnacipran, pregabalin, gabapentin, sodium oxybate or prohibited narcotics.
* Female patient who is pregnant, planning a pregnancy, or breastfeeding.
* Any anticipated need for surgery that might confound results or interfere with patient's ability to comply with the protocol.
* The occurrence of a major protocol violation during the lead-in study indicating a lack of compliance or other significant concern that precludes the patient's ongoing participation.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-08; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in patient 24-hour recall average pain intensity | Assessed at 12 weeks
  Pain intensity evaluated on a 100-mm visual analog scale (VAS)

SECONDARY OUTCOMES:
Patient self-reported Global Impression of Change | Assessed at 12 weeks
Change from baseline in Revised Fibromyalgia Impact Questionnaire | Assessed at 12 weeks
Change from baseline in patient 7-day recall average pain intensity | Assessed at 12 weeks
Change from baseline in Jenkins Sleep Questionnaire | Assessed at 12 weeks

OTHER OUTCOMES:
Change from baseline in Beck Depression Inventory (BDI-II) | Assessed at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Donald E Deering, PhD, Principal Investigator — St. Joseph Mercy Oakland; Jeffrey B Hargrove, PhD, Principal Investigator — Cerephex Corporation
Locations (1):
- St. Joseph Mercy Oakland, Pontiac, Michigan, United States

REFERENCES:
- [Background] Hargrove JB, Bennett RM, Simons DG, Smith SJ, Nagpal S, Deering DE. A randomized placebo-controlled study of noninvasive cortical electrostimulation in the treatment of fibromyalgia patients. Pain Med. 2012 Jan;13(1):115-24. doi: 10.1111/j.1526-4637.2011.01292.x. PMID 22233397
- [Background] Hargrove JB, Bennett RM, Clauw DJ. Long-term outcomes in fibromyalgia patients treated with noninvasive cortical electrostimulation. Arch Phys Med Rehabil. 2012 Oct;93(10):1868-71. doi: 10.1016/j.apmr.2012.04.006. Epub 2012 Apr 21. PMID 22525670